CLINICAL TRIAL: NCT05580835
Title: Added Value of PET / MR With PSMA for Diagnosis and Staging of Hepatocellular Carcinoma
Brief Title: PET / MR With PSMA for Diagnosis and Staging of Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Irai Santana de Oliveira, MD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 54382721.3.0000.0068
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Positron Emission Tomography/Magnetic Resonance) (PET/MR); Magnetic resonance imaging; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Patients with an imaging diagnosis of hepatocellular carcinoma and candidates to a liver transplant or surgical resection will be submitted to a novel imaging scan, PET / MRI with PSMA. The role of this imaging scan on diagnosis and staging of HCC will be evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PET MRI - PSMA (Experimental): Patients with an imaging diagnosis of HCC and submitted to PET MRI - PSMA
  Interventions: Diagnostic Test: PET MRI with PSMA

INTERVENTIONS:
Diagnostic Test: PET MRI with PSMA — A whole-body PET using PSMA as a radiotracer associated to an upper abdomen MRI with gadoxetic acid as contrast agent

SUMMARY:
Assess the rate and degree of PSMA uptake in patients with hepatocellular carcinoma submitted to PET/MRI scans. The objective is to evaluate its value on diagnosis and staging of HCC.

DETAILED DESCRIPTION:
PET/MR - PSMA have emerged as a new method and there are few studies about its role in the evaluation of hepatocellular carcinoma (HCC).

The hypothesis in this study is that PET/MRI with PSMA might have an additional value in the assessment of hepatocellular carcinoma, contributing to the diagnosis of distant metastasis and to confirm the diagnosis in undetermined nodules by the standard exams (computed tomography and magnetic resonance imaging).

Patients with hepatocellular carcinoma diagnosed by computed tomography or magnetic resonance imaging and referred to a liver transplant or surgery by clinical decision wil be submitted to a whole-body PSMA-PET/MRI and will be included in this prospective unicentric study to be conducted at Instituto do Câncer do Estado de São Paulo (ICESP) and Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HC-FMUSP).

All cases will be evaluated to determine the presence and degree of PSMA uptake on lesions considered as definitely HCCs by CT or MRI. The sensitivity of PSMA - PET/MR for the diagnosis of HCC will be calculated.

The added value of PSMA - PET MR on systemic staging will be calculated by the number of lesions considered suspicious for malignancy that were not detected by conventional scans.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an imaging diagnosis of HCC by a previous CT or MRI, reviewed by an abdominal radiologist
* Patients candidates to liver transplant or surgical resection

Exclusion Criteria:

* Patients with treated liver lesion without viable tumor
* Age under 18
* Pregnancy
* Patients with renal insufficiency;
* Elevated bilirubin levels (>3 mg/dL)
* Known allergy to contrast media (gadoxetic acid) or radiotracer (PSMA);
* Blood glucose level higher than 150 mg/dl.
* MR contraindications (claustrophobia, cardiac pacemakers, neurostimulators, cochlear implants, and insulin pumps).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-09-04 (Estimated); Study Completion 2024-09-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of PET MRI - PSMA for HCC | 24 months
  Patients with a liver lesion diagnosed as hepatocellular carcinoma by MRI or CT and candidates to surgical resection or liver transplant will be submitted to PET MRI with PSMA. Based on the presence or absence of PSMA uptake, sensitivity and specificity of PET MRI for diagnosis of the liver lesion and extrahepatic disease will be calculated.
Degree of PSMA uptake by HCC | 24 months
  For all liver lesions diagnosed as HCC, the degree of PSMA on PET uptake will be measured and correlated with available pathology information

SECONDARY OUTCOMES:
Correlation of PSMA uptake and liver nodules histology | 24 months
  All other non-HCC nodules simultaneously diagnosed will be also evaluated in terms of presence and degree of PSMA uptake. This results will be computed and correlated with all pathology data available
Presence of PSMA uptake on treated liver lesions | 24 months
  Whenever a treated observation is present, the presence and degree of PSMA uptake will be evaluated and correlated to conventional imaging scans and pathology results available

CONTACTS AND LOCATIONS:
Overall Officials: Irai S Oliveira, MD, Principal Investigator — University of Sao Paulo; Carlos Buchpiguel, PhD, Study Chair — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, Brazil